CLINICAL TRIAL: NCT04226157
Title: Home Blood Pressure Self-Management in Hypertensive Stroke Survivors: a Pilot Study
Brief Title: Home Blood Pressure Study for Recent Stroke Survivors With High Blood Pressure *On Hold Due to Global Pandemic*
Acronym: HBPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedStar Georgetown University Hospital (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Mary Carter Denny, Assistant Professor of Neurology, MedStar Georgetown University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0718
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Ischemic Stroke; Hypertension
Keywords: Blood Pressure; Stroke; Hypertension; Blood Pressure Monitor; Home Blood Pressure Monitor; Ischemic Stroke; Stroke Prevention
MeSH Terms: conditions — Ischemic Stroke; Hypertension; Stroke

STUDY DESIGN:
Intervention Model Description: Patients with hypertension who have had a stroke within the past 6 months will be randomized into two groups in a one to one ratio: Home Blood Pressure Self-Management (HBPS) or Usual Care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Blood Pressure Self Management (Experimental): The HBPS group will check their blood pressure at home daily using a smart BP cuff with telemonitoring capability (Home Qardio) and guided to use a self-titration plan between office visits for persistently elevate blood pressures.
  Interventions: Device: Home Blood Pressure Monitoring Device (Qardio Arm)
- Usual Care (Active Comparator): The Usual Care group will have their blood pressure monitored and medications adjusted by their primary care provider.
  Interventions: Other: Primary Care Provider Blood Pressure Management

INTERVENTIONS:
Device: Home Blood Pressure Monitoring Device (Qardio Arm) — The Home Blood Pressure Device with telemonitoring capability will allow the participants and physician to monitor blood pressure over time and titrate blood pressure medications as needed for persistently elevated blood pressure.
  Other Names: Medication Self-Titration
  Arms: Home Blood Pressure Self Management
Other: Primary Care Provider Blood Pressure Management — Participant will follow up as would normally do with primary care provider for blood pressure management.
  Arms: Usual Care

SUMMARY:
The purpose of this pilot study is to assess the feasibility of implementing a home blood pressure self-management program in a population of recent stroke survivors in the Washington, D.C. area. The investigators hypothesize that hypertensive stroke survivors in the Washington, DC area who participate in the Home Blood Pressure Monitoring program will have a greater reduction in mean systolic blood pressure (SBP) from baseline to 3 months, as measured by automated office blood pressure (AOBP), as compared to usual care.

DETAILED DESCRIPTION:
The purpose of this trial is to determine if a home blood pressure self-management (HBPS) program, including home monitoring and medication adjustments, is practical to use in recent stroke survivors and whether or not it is associated with lowering blood pressure after 3 months. Data from this trial may be used to do more research and may be used by doctors when seeing patients.This research is being done because high blood pressure, also called hypertension, is the leading risk factor for stroke. Lowering blood pressure (BP) has been shown to lower the risk of future strokes. The majority of stroke survivors continue to have uncontrolled BP. Currently, blood pressure (BP) is most often measured in the doctor's office. However, those single BP measurements are not the best picture of blood pressure over time and can be influenced by the stress of being in a doctor's office, known as the "white coat effect". This is why measuring BP at home may paint a more accurate picture of a patient's true long-term BP. Home blood pressure monitoring (HBPM) is recommended in the recently updated national hypertension guidelines. Home BP monitoring plus guided BP medication self-adjustments is associated with lower BP in patients with high blood pressure. The investigators believe that a HBPS program, including medication self-adjustment and home monitoring, may help to reduce blood pressure in patients with hypertension within 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke in the past 180 days of screening
* Age >/= 18 years old
* Automated Office Blood Pressure ≥135 systolic or ≥85 diastolic at time of screening
* Stage 2 hypertension (as defined by >140 mmHg SBP and or >90 mmHg DBP on 2 occasions or history of hypertension prior to stroke or currently taking antihypertensive medications)
* Able to live independently (as defined by modified Rankin scale score of 0-2)

Exclusion Criteria:

* CKD stage IV or greater (GFR < 30)
* Inability to check BP in either arm (e.g. amputation, lymphedema)
* Pregnancy
* High-grade intracranial or extracranial stenosis requiring a higher BP goal
* Unable to provide informed consent for themselves in English or Spanish
* Life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of blood pressure self management in stroke survivors | Three Months
  At least 75 percent of HBPS participants will successfully complete the monitoring and self-titration intervention.

SECONDARY OUTCOMES:
Systolic Blood Pressure Difference | three months
  Difference in systolic blood pressure from baseline to three months between HBPS and Usual Care arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ovbiagele B, Nguyen-Huynh MN. Stroke epidemiology: advancing our understanding of disease mechanism and therapy. Neurotherapeutics. 2011 Jul;8(3):319-29. doi: 10.1007/s13311-011-0053-1. PMID 21691873
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Petty GW, Brown RD Jr, Whisnant JP, Sicks JD, O'Fallon WM, Wiebers DO. Ischemic stroke subtypes : a population-based study of functional outcome, survival, and recurrence. Stroke. 2000 May;31(5):1062-8. doi: 10.1161/01.str.31.5.1062. PMID 10797166
- [Background] Katsanos AH, Filippatou A, Manios E, Deftereos S, Parissis J, Frogoudaki A, Vrettou AR, Ikonomidis I, Pikilidou M, Kargiotis O, Voumvourakis K, Alexandrov AW, Alexandrov AV, Tsivgoulis G. Blood Pressure Reduction and Secondary Stroke Prevention: A Systematic Review and Metaregression Analysis of Randomized Clinical Trials. Hypertension. 2017 Jan;69(1):171-179. doi: 10.1161/HYPERTENSIONAHA.116.08485. Epub 2016 Oct 31. PMID 27802419
- [Background] Law MR, Morris JK, Wald NJ. Use of blood pressure lowering drugs in the prevention of cardiovascular disease: meta-analysis of 147 randomised trials in the context of expectations from prospective epidemiological studies. BMJ. 2009 May 19;338:b1665. doi: 10.1136/bmj.b1665. PMID 19454737
- [Background] White CL, Pergola PE, Szychowski JM, Talbert R, Cervantes-Arriaga A, Clark HD, Del Brutto OH, Godoy IE, Hill MD, Pelegri A, Sussman CR, Taylor AA, Valdivia J, Anderson DC, Conwit R, Benavente OR; SPS3 Investigators. Blood pressure after recent stroke: baseline findings from the secondary prevention of small subcortical strokes trial. Am J Hypertens. 2013 Sep;26(9):1114-22. doi: 10.1093/ajh/hpt076. Epub 2013 Jun 4. PMID 23736109
- [Background] Hackam DG, Spence JD. Combining multiple approaches for the secondary prevention of vascular events after stroke: a quantitative modeling study. Stroke. 2007 Jun;38(6):1881-5. doi: 10.1161/STROKEAHA.106.475525. Epub 2007 Apr 12. PMID 17431209
- [Background] Lager KE, Mistri AK, Khunti K, Haunton VJ, Sett AK, Wilson AD. Interventions for improving modifiable risk factor control in the secondary prevention of stroke. Cochrane Database Syst Rev. 2014 May 2;(5):CD009103. doi: 10.1002/14651858.CD009103.pub2. PMID 24789063
- [Background] Siegel D. Barriers to and strategies for effective blood pressure control. Vasc Health Risk Manag. 2005;1(1):9-14. doi: 10.2147/vhrm.1.1.9.58940. PMID 17319093
- [Background] Berlowitz DR, Ash AS, Hickey EC, Friedman RH, Glickman M, Kader B, Moskowitz MA. Inadequate management of blood pressure in a hypertensive population. N Engl J Med. 1998 Dec 31;339(27):1957-63. doi: 10.1056/NEJM199812313392701. PMID 9869666
- [Background] Boden-Albala B, Quarles LW. Education strategies for stroke prevention. Stroke. 2013 Jun;44(6 Suppl 1):S48-51. doi: 10.1161/STROKEAHA.111.000396. No abstract available. PMID 23709728
- [Background] McManus RJ, Mant J, Haque MS, Bray EP, Bryan S, Greenfield SM, Jones MI, Jowett S, Little P, Penaloza C, Schwartz C, Shackleford H, Shovelton C, Varghese J, Williams B, Hobbs FD, Gooding T, Morrey I, Fisher C, Buckley D. Effect of self-monitoring and medication self-titration on systolic blood pressure in hypertensive patients at high risk of cardiovascular disease: the TASMIN-SR randomized clinical trial. JAMA. 2014 Aug 27;312(8):799-808. doi: 10.1001/jama.2014.10057. PMID 25157723
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Fernandez S, Chaplin W, Schoenthaler AM, Ogedegbe G. Revision and validation of the medication adherence self-efficacy scale (MASES) in hypertensive African Americans. J Behav Med. 2008 Dec;31(6):453-62. doi: 10.1007/s10865-008-9170-7. Epub 2008 Sep 11. PMID 18784996
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] de Man-van Ginkel JM, Hafsteinsdottir T, Lindeman E, Burger H, Grobbee D, Schuurmans M. An efficient way to detect poststroke depression by subsequent administration of a 9-item and a 2-item Patient Health Questionnaire. Stroke. 2012 Mar;43(3):854-6. doi: 10.1161/STROKEAHA.111.640276. Epub 2011 Dec 8. PMID 22156689